CLINICAL TRIAL: NCT01150162
Title: A Prospective Randomized, Multi-center Study to Assess the Safety and Efficacy of Mucosta (Rebamipide), in Combination With Omeprazole as Adjuvant Therapy in Gastric Ulcer Patients
Brief Title: Mucosta in Gastric Ulcer Treatment, Effectiveness and Safety Evaluation
Acronym: MGES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pakistan Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 037-POA-0901i
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Gastric Ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — rebamipide; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mucosta and Omeprazole (Experimental)
  Interventions: Drug: Rebamipide and Omeprazole
- Omeperazole (Active Comparator)
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Rebamipide and Omeprazole — open label, oral route, Rebamipide, 100mg tablet t.i.d and Omeprazole 20 mg tablet B.I.D. for 8 weeks
  Other Names: Mucosta; Omeprazole
  Arms: Mucosta and Omeprazole
Drug: Omeprazole — open label,oral route, Omeprazole 20mg tablet, B. I.D.; alone, for 8 weeks
  Arms: Omeperazole

SUMMARY:
A Prospective Randomized, Multi-center study to assess the Safety and Efficacy of Mucosta (Rebamipide), in combination with Omeprazole as adjuvant therapy in Gastric Ulcer Patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspepsia or epigastric pain and endoscopically proven gastric and duodenal ulcers
* Required laboratory parameters and time limits (screening blood tests will be taken including hemoglobin, white blood cell count, random glucose, potassium, sodium, chlorine, creatinine, AST, ALT, bilirubin, and alkaline phosphatase)
* Age > 18 years
* A statement that all patients must have signed an informed consent form prior to registration in study

Exclusion Criteria:

* Patients who had undergone surgery for ulcers
* History of hypersensitivity to drugs to be used in the study
* Women who are pregnant or lactating or intended to get pregnant during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Healing rates for gastric ulcer patients via endoscopic examination | 8 weeks treatment plus 4 weeks follow-up
Improvement or absence of gastric ulcer associated symptoms | 8 weeks treatment plus 4 weeks follow-up
  Improvement or absence of gastric ulcer associated symptoms, i.e. pain, burning, etc.

SECONDARY OUTCOMES:
To determine and compare the Safety profile in both the treatment arms. | 8 weeks treatment plus 4 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Laeeque Ahmed, Asst. Professor, Principal Investigator — Dr. Ziauddin University Hospital
Locations (3):
- Pakistan (3):
  - Abbasi Shaheed Hospital, Karachi
  - Dow University of Health Sciences, Karachi
  - Dr. Ziauddin University Hospital, Karachi